CLINICAL TRIAL: NCT05751473
Title: Reducing PTSD Symptoms in First Responders and Frontline Healthcare Workers Through Trauma-focused Treatment in Employee Assistance Programs
Brief Title: Reducing Posttraumatic Stress Disorder (PTSD) Symptoms in First Responders and Frontline Health Care Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Sripada, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00219260; 1R01MH126693-01 (NIH)
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Employee Assistance Programs; Frontline Healthcare Workers; Prolonged Exposure for Primary Care; First Responders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Primary Health Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Exposure for Primary Care (Experimental)
  Interventions: Behavioral: Prolonged Exposure for Primary Care (PE-PC)
- EAP Treatment as Usual (TAU) (Active Comparator): Employee Assistance Programs standard treatment.
  Interventions: Behavioral: EAP Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Prolonged Exposure for Primary Care (PE-PC) — Treatment will be given by telehealth or in person, depending on the participant preference.
  Content is drawn from the Full Prolonged Exposure model and condensed so as to deliver the most efficacious components in a brief format. There will be 4-6 weekly 30-minute sessions. Treatment follows the standardized PE-PC manual and workbook. At the end of the final session, the counselor and participant will review treatment progress and either conclude treatment or refer the participant to outside mental healthcare for more intensive treatment.
  Participants will complete surveys and complete homework during and following the study.
  Arms: Prolonged Exposure for Primary Care
Behavioral: EAP Treatment as Usual (TAU) — Treatment will be given by telehealth or in person, depending on the participant preference and current EAP practices (4-6 weeks). This will be the standard of care practice at each EAP site. Usually, this includes up to six sessions of solution focused therapy, and referrals to an established network of community providers who specialize in PTSD treatment. All PTSD care received during the study will be collected and monitored as TAU. The type of TAU used will reflect the current practice in EAPs and will not be constrained in the study design. EAP staff will monitor and record all EAP care received, including tracking no shows and cancellations. Study team members will document care received outside of the EAP (including psychiatric medications) by self-report.
  Participants will complete surveys and complete homework during and following the study.
  Arms: EAP Treatment as Usual (TAU)

SUMMARY:
This study addresses PTSD symptoms in First Responders and Healthcare workers. Specifically, it tests whether a brief PTSD treatment (talk therapy) effectively treats PTSD when provided to First Responders and Healthcare workers by counselors in Employee Assistance Programs (EAPs).

The central hypothesis is that the PTSD treatment, Prolonged Exposure for Primary Care (PE-PC), will reduce PTSD symptoms and improve functioning, compared to EAP Treatment as Usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Are employees at an orginization served by a participating EAP
* Have a Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) score ≥33
* Have had psychotropic medication stability for at least 4 weeks

Inclusion criteria for the qualitative portion of the study:

- Enrolled into the randomized clinical trial and were a treatment responder or were a treatment non-responder

Exclusion Criteria:

* Severe cognitive impairment that in the judgment of the investigators makes it unlikely that the participant can adhere to the study regimen (as evidenced by confusion, inability to track discussion or answer questions, or other clear and significant indicators of cognitive impairment)
* High risk of suicide (defined as meeting criteria for Action Step 3 on the Participant Suicide Risk Screening form: found in protocol)
* Need for detoxification
* Active psychosis or unmanaged bipolar disorder, as measured by items 12 and 13 of the cross cutting assessment
* Currently engagement in a trauma-focused behavioral treatment (such as Prolonged Exposure or Cognitive Processing Therapy).
* Patients who do not speak English will be excluded for logistical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) score | baseline to 6 months
  The PCL-5 is a 20-item self-report measure that assesses symptoms of PTSD. The self-report rating scale is 0-4 for each symptom. The minimum and maximum values are 0 and 80, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Change in Burnout based on the Oldenburg Burnout Inventory | baseline to 6 months
  This is a 16-question inventory that assesses burnout. The self-report rating scale is 1-4 for each symptom.The minimum and maximum values are 16 and 64, with higher scores indicating worse outcome.
Change in Job Performance based on the Work Productivity and Activity Impairment Questionnaire (WPAI-GH) | baseline to 6 months
  The WPAI-GH measures the impact of health problems on absenteeism, presenteeism, overall work performance and non-work activities using a 0 to 10 visual analog scale (VAS).
Change in Depressive Symptoms based on the Patient Health Questionnaire (PHQ-9) | baseline to 6 months
  This is a 9-item questionnaire that participants select responses from not at all (0) to nearly every day (3), the minimum and maximum score values ranging from 0 to 27. Higher scores indicate a worse outcome and lower scores indicate better outcome.
Change in Patient Satisfaction based on the Client Satisfaction Questionnaire (CSQ-8) | baseline to 6 months
  This is an 8-item questionnaire that participants complete. Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sripada, PhD, Principal Investigator — University of Michigan
Locations (12):
- United States (12):
  - Sharp Healthcare, San Diego, California
  - Tanner Health System, Carrollton, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Detroit Fire Department, Detroit, Michigan
  - Health Management Systems of America, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - West Bloomfield Fire Department, West Bloomfield, Michigan
  - Cope NewYork-Presbyterian, New York, New York
  - University of Cincinati Health, Cincinnati, Ohio
  - ProMedica, Fremont, Ohio
  - Houston Fire Department, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sripada RK, Garlick J, Hemphill N, Walters HM, Ganoczy D, Kim HM, Zivin K, Nevedal AL, Avallone KM, Cigrang JA, Rauch SAM. Addressing PTSD symptoms in first responders and healthcare workers through trauma-focused treatment in Employee Assistance Programs: Protocol for a randomized controlled trial. Contemp Clin Trials. 2026 Jan;160:108174. doi: 10.1016/j.cct.2025.108174. Epub 2025 Dec 4. PMID 41352531